CLINICAL TRIAL: NCT04941521
Title: Feasibility of Exenatide, a GLP-1R Agonist, for Treating Cocaine Use Disorder: A Case Series Study
Brief Title: Exenatide for Treating Cocaine Use Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Joy Schmitz, Professor, Faillace Chair, and Director for the Center for Neurobehavioral Research on Addiction, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-21-0241
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Results first posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-03

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine use; Exenatide; Cocaine treatment
MeSH Terms: interventions — Exenatide

STUDY DESIGN:
Intervention Model Description: Case series design run as a single-arm open-label pilot
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Exenatide and Drug Counseling (Experimental): Participants will receive once weekly exenatide injections and drug counseling sessions.
  Interventions: Drug: Exenatide 2 mg [Bydureon]; Behavioral: Drug Counseling

INTERVENTIONS:
Drug: Exenatide 2 mg [Bydureon] — Exenatide will be purchased commercially as Bydureon® for subcutaneous (SC) injection and administered at a dose of 2 mg once a week for a total of 6 weeks. Each single-dose, dual-chamber pen contains 0.65 mg of diluent and 2 mg of exenatide, which remains isolated until mixed.
  Other Names: Bydureon
Behavioral: Drug Counseling — Once weekly drug counseling sessions for cocaine use with trained masters-level therapists.

SUMMARY:
The purpose of this study is to collect information about whether exenatide (Bydureon) may be safe and helpful as a medication treatment for individuals who want to stop using cocaine.

Although exenatide (Bydureon) is approved by the Food and Drug Administration (FDA) for the treatment of type 2 diabetes, it has not been approved by the FDA to treat cocaine use; therefore, it is called an investigational drug.

DETAILED DESCRIPTION:
Cocaine use continues to be a significant public health problem with limited treatment options and no approved pharmacotherapies. Glucagon-like peptide 1 (GLP-1) receptors are located in brain areas important for reward and, as such, appear to play a significant role in modulating addictive-like behaviors and drug use (Eren-Yazicioglu et al. 2020). Extended-release exenatide is a GLP-1 receptor agonist approved by the FDA for the treatment of type 2 diabetes. In preclinical studies, exenatide reduces cocaine-seeking and cocaine-taking behavior (Brunchmann et al. 2019). The effect of extended-release exenatide on cocaine use in patients with a cocaine use disorder (CUD) has not yet been investigated. A series of four case studies are being proposed to collect preliminary data on the feasibility, safety, and clinical effects of exenatide in treatment-seeking patients with CUD.

The U.S. is facing a re-emergence of cocaine as an epidemic drug, indicated by increases in availability, use, and overdose deaths following a previous period of decline (Maxwell 2020). Although significant strides have been made in medication development for the treatment of cocaine use disorder (CUD), no FDA-approved pharmacotherapies are currently available. NIDA's current strategic plan prioritizes efforts to accelerate CUD medication development by rigorously testing novel molecular targets based on a translational research approach. Emerging evidence supports the potential clinical utility of glucagon-like peptide 1 (GLP-1) receptor stimulation for the treatment of substance use disorders, including CUD.

GLP-1 is an incretin hormone that promotes insulin secretion from pancreatic beta cells. Current evidence shows that GLP-1 receptors are widely expressed in areas of the mesolimbic dopaminergic pathway where they regulate the rewarding value of food and drugs of abuse, including cocaine. Preclinical literature suggests that activation of GLP-1 receptors reduces the rewarding effects of cocaine and cocaine self-administration (e.g., Hernandez et al. 2018; Hernandez et al. 2019). In the human laboratory, acute cocaine administration decreases GLP-1 concentrations, with changes associated with subjective reinforcing responses to cocaine ("feeling high, anxious") (Bouhlal et al. 2017). Thus, there is compelling evidence to hypothesize that exenatide treatment will decrease cocaine use in individuals with CUD. In preparation for conducting a full-scale efficacy trial, the goal of the current proposal is to collect preliminary feasibility, safety, and clinical data on the effects of exenatide in series of four case studies.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 60 years of age.
* meet DSM-5 criteria for current cocaine use disorder as measured by the Structured Clinical Interview for DSM-5 (SCID).
* have at least 1 cocaine-positive urine specimen (≥ 150 ng/mL) during intake.
* be in acceptable health on the basis of interview, medical history and physical exam.
* have hematology and chemistry laboratory tests that are within reference limits (±10%), with the following exception: pancreatic tests (lipase and amylase) must be within normal limits.
* consent to use an acceptable method of birth control during study participation and for one month after discontinuation of the study medication. Non-hormonal methods of contraception are recommended, including barrier contraceptives (e.g., diaphragm, cervical cap, male condom) or intrauterine device (IUD). Steroid contraceptives if used with non-hormonal methods are acceptable.
* be able to understand the consent form and provide written informed consent.
* be able to provide the names of at least 2 persons who can generally locate their whereabouts.

Exclusion Criteria:

* current DSM-5 diagnosis for substance use disorder (of at least moderate severity) other than cocaine, marijuana, alcohol, or nicotine.
* current alcohol use that meets for physiological dependence requiring detoxification or makes participation medically unsafe as determined by the medical director.
* have a DSM-5 axis I psychiatric disorder, or anorexia nervosa, or neurological disease or disorder requiring ongoing treatment and/or making study participation unsafe (e.g., psychosis, dementia).
* significant current suicidal or homicidal ideation.
* Type 1 or type 2 diabetes mellitus (previously diagnosed or indicated by HbA1C level of ≥6.5%).
* have medical conditions contraindicating exenatide pharmacotherapy (e.g., personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2, severe gastrointestinal disease (severe gastroparesis), previous history of pancreatitis or risk of pancreatitis, creatinine clearance <45 or end stage renal disease, previous medically adverse reaction to exenatide or other GLP-1 receptor agonists).
* taking medications that could adversely interact with exenatide (e.g., oral or injectable blood glucose lowering medications).
* having conditions of probation or parole requiring reports of drug use to officers of the court.
* impending incarceration.
* pregnant or nursing for female patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy Schmitz, PhD, Principal Investigator — UT Houston; Luba Yammine, PhD, Principal Investigator — UT Houston
Locations (1):
- UTHealth Behavioral and Biomedical Sciences Building, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers.

REFERENCES:
- [Derived] Yammine L, Balderas JC, Weaver MF, Schmitz JM. Feasibility of Exenatide, a GLP-1R Agonist, for Treating Cocaine Use Disorder: A Case Series Study. J Addict Med. 2023 Jul-Aug 01;17(4):481-484. doi: 10.1097/ADM.0000000000001147. Epub 2023 Feb 17. PMID 37579116

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exenatide and Drug Counseling
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.33 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
Number of Years of Education [Mean (Standard Deviation); unit: years] | 13.00 (3.60)
Tobacco Dependency assessed by the Fagerstrom Test [Count of Participants; unit: Participants] — Tobacco dependence was assessed by the Fagerstrom Test for Nicotine Dependence, and results are reported categorically from very low dependence to very high dependence.
  Participants
    Very Low Dependence | 1
    Low Dependence | 0
    Medium Dependence | 1
    High Dependence | 1
    Very High Dependence | 0
number of days of use of cocaine in the past 30 days [Mean (Standard Deviation); unit: days] | 18 (7)
number of days use of alcohol in the past 30 days [Mean (Standard Deviation); unit: days] | 8 (5.29)
number of days use of marijuana in the past 30 days [Mean (Standard Deviation); unit: days] | 8.33 (10.21)
number of years use of cocaine [Mean (Standard Deviation); unit: years] | 17 (13.52)
number of years use of alcohol [Mean (Standard Deviation); unit: years] | 9.33 (8.38)
number of years use of Marijuana [Mean (Standard Deviation); unit: years] | 3.33 (5.77)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by Number of Participants Who Completed Treatment
Description: Treatment completion will be assessed by attendance at the end-of-treatment timepoint.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Drug Safety as Assessed by Total Number of Adverse Events Reported During Treatment
Description: Adverse events (AEs) will be reported to study nurse during the course of treatment.
Time Frame: From Week 1 to Week 6
Measure: Number; unit: adverse events
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
adverse events | 7

3. Primary Outcome: Clinical Effect of Exenatide as Assessed by Cocaine Use During Treatment as Indicated by Number of Participants With Cocaine-positive Urine Drug Screen Results
Description: Urine drug screens were performed weekly. For a cocaine-negative urine drug screen result, benzoylecgonine levels must be under 300 ng/mL.
Time Frame: From Week 1 to Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
Participants
  week 1 | 3
  week 2 | 3
  week 3 | 3
  week 4 | 2
  week 5 | 2
  week 6 | 2

4. Secondary Outcome: Feasibility as Assessed by Number of Participants Enrolled
Description: Enrollment will be assessed by the number of participants signing the informed consent.
Time Frame: Week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
Participants | 3

5. Secondary Outcome: Feasibility as Assessed by Number of Study Visits Attended
Description: There were 6 study visits planned.
Time Frame: From Week 1 to Week 6
Measure: Mean (Standard Deviation); unit: study visits
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
study visits | 6 (0)

6. Secondary Outcome: Feasibility as Assessed by Retention as Indicated by Total Number of Completed Study Visits
Description: Retention will be assessed by the total number of completed study visits. A completed study visit is a visit in which the participant attended and received the study treatment.
Time Frame: From Week 1 to Week 6
Measure: Mean (Standard Deviation); unit: completed study visits
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
completed study visits | 6 (0)

7. Secondary Outcome: Feasibility as Indicated by Overall Acceptability as Reported on the Satisfaction Survey
Description: The Satisfaction Survey includes a 9-point likert scale that ranges from 1 to 9, with a higher score indicating greater acceptability.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
score on a scale
  treatment helpfulness | 7.66 (1.52)
  treatment usefulness | 6.00 (3.00)
  likelihood of treatment recommendation | 7.33 (2.88)
  desire to continue treatment | 7.33 (2.08)

8. Secondary Outcome: Clinical Effect of Exenatide as Assessed by Number of Participants Who Self-reported Cocaine Use on 50% or More Days of the Week
Description: Timeline Followback (TLFB) administered once weekly.
Time Frame: From Week 1 to Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
Participants
  week 1 | 2
  week 2 | 2
  week 3 | 1
  week 4 | 2
  week 5 | 1
  week 6 | 2

9. Secondary Outcome: Clinical Effect of Exenatide as Indicated by Number of Participants Who Reported a Reduction in Craving by Week 6 as Indicated by Cocaine Craving on the Brief Substance Craving Scale
Description: The brief substance craving scale (BSCS) is a 16-item, self-report instrument that assesses craving for cocaine and other substances of abuse over a 24 hour period. The domains of intensity, frequency, and duration are recorded on a five-point Likert scale. The range of scores for each domain is 0 to 4, and the total score is the sum of all three domains. The total score range is 0 to 12, and higher scores indicate higher craving (worse outcome.)
Time Frame: From Week 0 to Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
Participants | 2

10. Secondary Outcome: Clinical Effect of Exenatide as Assessed by Number of Participants Who Had a Decrease in Drug Demand by Week 6
Description: Drug demand will be measured by the computerized Cocaine Purchasing Task (CPT). The CPT asks participants how much cocaine they would purchase at the beginning of a hypothetical day as the cost of cocaine increases from $0 to $1,000. The CPT simulates changes in price and consumption of drug in order to assess demand curves associated with drug consumption. The CPT will assess both cocaine reward value as well as motivation to consume cocaine.
Time Frame: From Week 0 to Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
Participants | 1

11. Secondary Outcome: Clinical Effect of Exenatide as Assessed by Number of Participants Who Were Below the Clinical Range for Depression by Week 6 as Indicated by the Beck Depression Inventory
Description: The Beck Depression Inventory score ranges from 0 to 63, with a higher score indicating greater depressive symptoms. The scores from each timepoint will be plotted as a trend line.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
Participants | 3

12. Secondary Outcome: Clinical Effect of Exenatide as Indicated by Number of Participants Who Had an Increase in Positive Affect Symptoms by Week 6 as Indicated on the Positive/Negative Affect Schedule
Description: The Positive/Negative Affect Schedule is a 20-item questionnaire divided into 10 positive affect items and 10 negative affect items. The score for the positive affect items ranges from 10 to 50, with a higher score indicating higher levels of positive affect. The scores from each timepoint will be plotted as a trend line.
Time Frame: From Week 0 to Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
Participants | 1

13. Secondary Outcome: Clinical Effect of Exenatide as Indicated by Number of Participants Who Had a Decrease in Negative Affect Symptoms Indicated on the Positive/Negative Affect Schedule
Description: The Positive/Negative Affect Schedule is a 20-item questionnaire divided into 10 positive affect items and 10 negative affect items. The score for the negative affect items ranges from 10 to 50, with a lower score indicating lower levels of negative affect. The scores from each timepoint will be plotted as a trend line.
Time Frame: From Week 0 to Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide and Drug Counseling
Number analyzed (Participants) | 3
Participants | 1

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Exenatide and Drug Counseling
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide and Drug Counseling (N=3)
Chest pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide and Drug Counseling (N=3)
Nausea (General disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Headache (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Injection Site Pruritus (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT04941521/Prot_SAP_000.pdf